CLINICAL TRIAL: NCT01054768
Title: Antioxidant Therapy to Reduce Inflammation in Sickle Cell Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009-003; 1R21AT004493-01 (NIH)
Record Dates: First submitted 2010-01-20; First posted 2010-01-22 (Estimated); Results first posted 2021-08-03 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Anemia, Sickle Cell
Keywords: Antioxidant; Inflammation; Sickle Cell Disease; Oxidative Stress; Cytokines; anti-inflammatory; Acetylcarnitine
MeSH Terms: conditions — Anemia, Sickle Cell; Inflammation | interventions — Thioctic Acid; Acetylcarnitine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- alpha-lipoic acid and acetyl-L-carnitine (Experimental): alpha-lipoic acid and acetyl-L-carnitine1400 mg tablet twice a day for 6 months.
  Interventions: Drug: alpha-lipoic acid and acetyl-L-carnitine
- Placebo (Placebo Comparator): 1400 mg placebo tablet twice a day for 6 months.
  Interventions: Drug: Control

INTERVENTIONS:
Drug: alpha-lipoic acid and acetyl-L-carnitine — none to report
  Other Names: Experimental
  Arms: alpha-lipoic acid and acetyl-L-carnitine
Drug: Control — none to report
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether alpha-lipoic acid and acetyl-L-carnitine will lower systemic inflammation in patients with Sickle Cell Disease by reducing oxidative stress, which will result in a decrease in the frequency of vaso-occlusive pain episodes and improve their quality of life.

DETAILED DESCRIPTION:
People with sickle cell disease have more inflammation (a response of body tissues to injury or irritation) than people without sickle cell disease. This inflammation can be measured in the blood by checking the level of a protein called C reactive protein as well as other changes we see in blood due to inflammation (such as changes in platelets and other cells). There is even more inflammation during sickle-related complications (like pain or acute chest syndrome). We want to test if inflammation in people with sickle cell disease can be reduced by the use of antioxidant compounds.

Antioxidants are nutrients (certain vitamins, minerals and enzymes) that can counteract the effects of oxidative stress arising from free radicals in our cells. The formation of free radicals is a normal cell process, but uncontrolled oxidative stress can cause problems for us. One such harmful problem is inflammation.

We know from other research studies that antioxidants help with some conditions related to inflammation. In this study the antioxidant being tested is a combination of alpha-lipoic acid and acetyl-L-carnitine, both of which are natural parts of many of the foods we eat and are needed by our cells to make energy from food.

ELIGIBILITY:
Inclusion Criteria:

* Proven diagnosis of sickle cell disease, either homozygous sickle disease or Hb S Beta zero thalassemia genotype
* Age at entry at least 14 years. Younger children will not be included since the combination alpha-lipoic acid and acetyl-L-carnitine tablets are not available in a smaller dose at this time.

Exclusion Criteria:

* More than 3 packed red blood transfusions in the past 12 months
* Coexisting illness that could contribute to inflammation. These include chronic hepatitis, lupus, arthritis, inflammatory bowel disease, chronic osteomyelitis, and other similar conditions.
* Acute sickle cell disease related symptoms requiring a hospital visit in the past 4 weeks
* Women who are pregnant, attempting to get pregnant, or breast feeding
* Active participation in other investigational drug or device studies
* Participants who start hydroxyurea or regular transfusion therapy during the course of the study on the recommendation of their primary hematologist will be ineligible for further participation.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2009-08; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elliott Vichinsky, M.D., Principal Investigator — UCSF Benioff Children's Hospital Oakland; Bruce N. Ames, Ph.D., Study Chair — UCSF Benioff Children's Hospital Oakland; Ashutosh Lal, M.D., Study Director — UCSF Benioff Children's Hospital Oakland
Locations (1):
- Children's Hospital & Research Center Oakland, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject was enrolled 08/10/09. Length of subject involvement was 7 months. Each subject was seen once a month at Children's Hospital & Research Center Oakland
Pre-assignment Details: Exclusions included those with 3 packed red blood transfusions in the past year, illness that could contribute to inflammation, acute sickle cell disease related symptoms requiring a hospital visit, those pregnant or breast feeding, or in other investigational drug or device studies, participants on hydroxyurea or a regular transfusion therapy.
Groups:
- Alpha-lipoic Acid and Acetyl-L-carnitine: alpha-lipoic acid and acetyl-L-carnitine 1400 mg tablet twice a day for 6 months.
  alpha-lipoic acid and acetyl-L-carnitine: none to report
- Placebo: 1400 mg placebo tablet twice a day for 6 months.
  Placebo: none to report
Period: Overall Study
Arm/Group | Alpha-lipoic Acid and Acetyl-L-carnitine | Placebo
Started | 17 | 20
Completed | 9 | 17
Not Completed | 8 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alpha-lipoic Acid and Acetyl-L-carnitine | Placebo | Total
Number analyzed (Participants) | 17 | 20 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 4 | 5
  Between 18 and 65 years | 16 | 16 | 32
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 10 | 12 | 22

OUTCOME MEASURES:

1. Primary Outcome: C-Reactive Protein
Description: C-Reactive Protein (CRP) was measured by a clinical laboratory. Measuring the quantity of serum CRP is helpful in recognizing inflammatory states.
Time Frame: 6 months
Population: Reason for discontinuation: started transfusions (2), alternative treatment (2), adverse events (4), subject preference (3).
Measure: Mean (Standard Deviation); unit: mg/l
Arm/Group | Alpha-lipoic Acid and Acetyl-L-carnitine | Placebo
Number analyzed (Participants) | 9 | 17
mg/l | 11.4 (20.9) | 6.8 (10.3)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Alpha-lipoic Acid and Acetyl-L-carnitine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/20
Serious Adverse Events (participants affected / at risk) | 8/17 | 9/20
Other Adverse Events (participants affected / at risk) | 6/17 | 12/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alpha-lipoic Acid and Acetyl-L-carnitine (N=17) | Placebo (N=20)
Vaso-occlusive pain (Blood and lymphatic system disorders) | 6 (13) | 9 (13)
Pneumonia/Acute Chest Syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alpha-lipoic Acid and Acetyl-L-carnitine (N=17) | Placebo (N=20)
Respiratory Symptoms (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 9 (12)
Nausea (Gastrointestinal disorders) | 2 (2) | 7 (7)
Urinary Urgency/UTI (Renal and urinary disorders) | 2 (2) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes